

### Statistical Analysis Plan

NCT Number: NCT05020015

an icable terms of Use applicable terms of Use applicable terms of Use Title: A Phase 2, Open-label, Multicenter Study of the Safety and Efficacy of TAK-007 in Adult Patients With Relapsed or Refractory B-cell Non-Hodgkin Lymphoma

Study Number: TAK-007-2001

Document Version and Date: Version 2.0, 30 Aug 2024

Certain information within this document has been redacted (ie, specific content is masked irreversibly from view) to protect either personally identifiable information or company

Property of Takeda. For noncommercial use only and property of Takeda.



## STATISTICAL ANALYSIS PLAN

Study Number: TAK-007-2001

A Phase 2, Open-label, Multicenter Study of the Safety and Efficacy of TAK-007 in Adult Patients With Relapsed or Refractory B-cell Non-Hodgkin Lymphoma

Phase: 2

Version: 2.0

Date: 30 August 2024 ...)
, Oncology SQS

Prepared by:

, PhD

Based on:

Protocol Version: Amendment 5 Protocol Date: 03 June 2024

#### CONFIDENTIAL PROPERTY OF TAKEDA

This document is a confidential communication of Takeda. Acceptance of this document constitutes the agreement by the recipient that no information contained herein will be published or disclosed without written authorization from Takeda.

#### **REVISION HISTORY**

| Version | Approval Date | Primary Rationale for Revision |
|---|---|---|
| Original | 09-Aug-2021 | Primary Rationale for Revision [Not Applicable] |
| Amendment 1 | | To make SAP consistent with Amendment 5 of the protocol, removal of Part 2 from the study |
| ity of Lakeda. | Fornonicommer | To make SAP consistent with Amendment 5 of the protocol, removal of Part 2 from the study |

# **TABLE OF CONTENTS**

| 1.0 | | OBJEC | CTIVES AND ENDPOINTS | 8 |
|---|---|---|---|---|
| | 1.1 | | jectives | |
| | | 1.1.1 | Primary Objectives | ~S.8 |
| | | 1.1.2 | Secondary Objectives | 8 |
| | | 1.1.3 | Exploratory Objectives | 8 |
| | 1.2 | En | Exploratory Objectives dpoints Primary Endpoints Secondary Endpoint(s) Exploratory Endpoint(s) Y DESIGN ISTICAL HYPOTHESES AND DECISION RULES | 8 |
| | | 1.2.1 | Primary Endpoints | 8 |
| | | 1.2.2 | Secondary Endpoint(s) | 8 |
| | | 1.2.3 | Exploratory Endpoint(s) | 9 |
| 2.0 | | STUD | Y DESIGN | 9 |
| 3.0 | | STATI | STICAL HYPOTHESES AND DECISION RULES | 10 |
| | 3.1 | Sta | itistical Hypotheses | 10 |
| | 3.2 | Mu | ultiplicity Adjustment | 10 |
| 4.0 | | SAMP | ttistical Hypotheses Iltiplicity Adjustment LE-SIZE DETERMINATION YSIS SETS ent-to-treat (ITT) set | 10 |
| 5.0 | | ANAL | YSIS SETS | 10 |
| | 5.1 | Inte | ent-to-treat (ITT) set | 10 |
| | 5.2 | Saf | fety analysis and Modified Intent-to-treat (mITT) set | 10 |
| | 5.3 | Res | sponse-evaluable analysis set | 10 |
| | 5.4 | CK | analysis setarmacodynamic analysis set | 10 |
| | 5.5 | Pha | armacodynamic analysis set | 10 |
| | 5.6 | Per | r-Protocol (PP) set | 11 |
| 6.0 | | | STICAL ANALYSIS | |
| | 6.1 | Ge | neral Considerations | |
| | | 6.1.1 | Definition of Study Visit Windows | |
| | | 6.1.2 | Conventions for Missing/Partial Dates in Screening Visit | |
| | | 6.1.3 | Conventions for Partial or Missing Adverse Event Dates | |
| | | | Conventions for Missing Concomitant Medication/Therapy Dates | 13 |
| | Ŏ | 6.1.5 | Conventions for Partial or Missing Subsequent Medication/Therapy Dates | 13 |
| X | 4. | 6.1.6 | Conventions for Partial or Missing Death Dates | |
| 50. | 6.2 | | sposition of Subjects | |
| | 6.3 | De | mographic and Other Baseline Characteristics | |
| | | 6.3.1 | Demographics and Baseline Characteristics | |
| | 6.4 | | edical History and Concomitant Medications | 15 |
| | 6.5 | A n | y Prior Interventions | 1.5 |

| 6.5.1 | Prior Anti-cancer Therapy | 15 |
|---|---|---|
| 6.5.2 | Other Prior Interventions | 15 |
| 6.6 E | Efficacy Analysis | 16 |
| 6.6.1 | Primary Endpoint Analysis | <u>.</u> 6 |
| 6.6.2 | Secondary Efficacy Endpoint(s) Analysis | 16 |
| 6 | 5.6.2.1 ORR by Investigator | 16 |
| 6 | 5.6.2.2 CR by Investigator | 16 |
| 6 | Primary Endpoint Analysis | 16 |
| 6 | 5.6.2.4 PFS by Investigator | 18 |
| 6 | 0.6.2.5 OS@ | 18 |
| 6.6.3 | Subgroup Analyses | 18 |
| 6.7 S | Safety Analysis | 20 |
| 6.7.1 | Adverse Events | 20 |
| 6.7.2 | Adverse Events of Clinical Interest | 21 |
| 6.7.3 | Other Safety Analysis | 22 |
| 6.7.4 | Extent of Exposure and Compliance | 22 |
| 6.8 C | CK, Pharmacodynamic, and Other Artalyses | 22 |
| 6.8.1 | CK Analyses | 22 |
| 6.8.2 | CK Analyses Pharmacodynamic Analyses | 24 |
| 6.9 In | mmunogenicity Analyses | 24 |
| 6.10 R | mmunogenicity Analyses RCR Analyses Exploratory Analyses | 24 |
| 6.11 E | Exploratory Analyses | 24 |
| 6.11. | | 24 |
| 6.11. | | |
| 6.11. | .3 Imaging Analyses | 25 |
| 6.11. | .4 PRO Analyses | 25 |
| 6.11, | 5 Healthcare Resource Utilization Analyses | 25 |
| | Statistical Considerations for Dose Escalation | |
| 6.13 In | nterim Analysis and Criteria for Early Termination | |
| 6.14 D<br>0 REFI | Data Monitoring Committee | 26 |
| 0 REF | ERENCES | 26 |
| | NGES TO PROTOCOL PLANNED ANALYSES | |
| 0 APPI | FNDIX | 27 |

#### LIST OF IN-TEXT TABLES

| Table 4 Dose Escalation/De-escala | tion Rule for the BOIN Design |
|---|---|
| | ssments and Censoring for DOR Primary Analysis |
| | , use only and |
| n.com | lercial de la company de la co |
| regs; ko, vo, | |
| et sie | |

#### ABBREVIATIONS

ΑE

AECI

area under the concentration-time curve from time 0 to time of the last quantifiable concentration
below the limit of quantification

Bayesian and the second secon  $AUC_{last}$ 

**BLO** BOIN Bayesian optimal interval CAR chimeric antigen receptor CI confidence interval

CK cellular kinetic(s)

Clast last measurable concentration maximum observed concentration  $C_{max}$ 

CR complete response

**CRS** cytokine release syndrome **CSR** clinical study report CTcomputed tomography

Common Terminology Criteria for Adverse Events **CTCAE** 

CV% percent coefficient of variation

Droplet Digital Polymerase Chain Reaction ddPCR

diffuse large B-cell lymphoma **DLBCL** 

DLT dose-limiting toxicity

DOB date of birth

**DOR** duration of response **DMC Data Monitoring Committee** 

**ECOG** Eastern Cooperative Oncology Group

ЕСНО echocardiogram

European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire EORTC-

QLQ-C30

European Quality of Life 5-Dimension 5-Level Scale EQ-5D-5L FACT-GP5 Functional Assessment of Cancer Therapy – General <sup>18</sup>F-fluorodeoxyglucose–positron emission tomography **FDG-PET** 

FL follicular lymphoma

**FLIPI** Follicular lymphoma international prognostic index

GvHD graft-versus-host disease HLA anti-human leukocyte antigen

**I**ČANS immune effector cell-associated neurotoxicity syndrome

ILinterleukin

iNHL indolent non-Hodgkin lymphoma

IPI international prognostic index for diffuse large B-cell lymphoma

intention-to-treat ITT

**IRC** Independent Review Committee

| | LBCL | large B-cell lymphoma |
|---|---|---|
| | LDH | Lactate dehydrogenase |
| | mAb | monoclonal antibody |
| | MedDRA | Medical Dictionary for Regulatory Activities |
| | mITT | modified intent to treat |
| | MRI | magnetic resonance imaging |
| | MZL | marginal zone lymphoma |
| | NCI | National Cancer Institute |
| | NHL | non-Hodgkin Lymphoma |
| | NK | natural killer (cells) |
| | ORR | overall response rate |
| | OS | overall survival |
| | PD | progressive disease |
| | PFS | progression free survival |
| | PP | per-protocol analysis set |
| | PR | partial response |
| | PT | Preferred Term (MedDRA) |
| | Q1 | monoclonal antibody Medical Dictionary for Regulatory Activities modified intent to treat magnetic resonance imaging marginal zone lymphoma National Cancer Institute non-Hodgkin Lymphoma natural killer (cells) overall response rate overall survival progressive disease progression free survival per-protocol analysis set partial response Preferred Term (MedDRA) 25th percentile 75th percentile relapsed or refractory replication competent retrovirus recommended phase 2 dose |
| | Q3 | 75th percentile |
| | r/r | relapsed or refractory |
| | RCR | replication competent retrovirus |
| | RP2D | recommended phase 2 dose |
| | SAE | serious adverse event |
| | SAP | statistical analysis plan |
| | SCT | stem cell transplantation |
| | SD | standard deviation |
| | TEAE | treatment-emergent adverse event |
| | | ·× |
| | · No | |
| | 67.0 | |
| | , 0 | |
| | les, | |
| | -0 <sup>©</sup> , | |
| | 101 | |
| X | TEAE TEAE | |

#### 1.0 OBJECTIVES AND ENDPOINTS

# 1.1 Objectives

#### 1.1.1 Primary Objectives

• To evaluate the safety and tolerability of TAK-007 in adult patients with relapsed or refractory (r/r) B-cell non-Hodgkin lymphoma (NHL) to determine the recommended phase 2 dose (RP2D).

## 1.1.2 Secondary Objectives

- To evaluate secondary efficacy endpoints (overall response rate (ORR), complete response [CR], duration of response [DOR], progression-free survival [PFS], and overall survival [OS]).
- To further evaluate the safety and tolerability of TAK-007 in adult patients with r/r large B-cell lymphoma (LBCL) and indolent non-Hodgkin lymphoma (iNHL).
- To characterize cellular kinetics (CK) of TAK-007.
- To assess pharmacodynamics of TAK-007.
- To assess immunogenicity of TAK-007

#### 1.1.3 Exploratory Objectives

- To conduct CK/pharmacodynamics modeling to further evaluate the relationship between exposure and response (safety, efficacy, pharmacodynamics, and product attributes).
- To explore biomarkers of clinical response including predictive biomarkers, mechanism of action, mechanism of resistance, and product performance.

#### 1.2 Endpoints

#### 1.2.1 Primary Endpoints

• Incidence of adverse events (AEs) and clinically significant laboratory values and vital signs.

# 1.2.2 Secondary Endpoints

- ORR per investigator.
- CR investigator.
- DOR investigator.
- PFS investigator.
- OS.

- CK parameters (eg, maximum observed concentration [C<sub>max</sub>], time of first occurrence of C<sub>max</sub> [t<sub>max</sub>], persistence (time of last measurable concentration above the lower limit of quantitation [t<sub>last</sub>]), area under the concentration-time curve from time 0 to time of the last quantifiable concentration [AUC<sub>last</sub>]), and other parameters as appropriate.
- Pharmacodynamic biomarker assessments utilizing B cell quantification and levels of cytokines in circulation over time.
- Prevalence and incidence of antidrug antibodies (ie, anti-human leukocyte antigen [HLA], anti-CAR).
- Prevalence and incidence of replication competent retrovirus (RCR) positive test results.

## 1.2.3 Exploratory Endpoints

- Characterization and evaluation of predictive biomarkers, as well as molecular mechanisms of action and resistance to TAK-007 utilizing (including but not limited to) quantitative and phenotypic evaluation of immune cells and cellular product characteristics, as well as HLA and KIR characterization.
- Assessment of circulating tumor DNA (ctDNA)
- Assessment of standardized uptake value, metabolic tumor volume, tumor volume computed tomography (CT)/magnetic resonance imaging (MRI), volumetric tumor assessment, and total lesion glycolysis assessed by <sup>18</sup>F-fluorodeoxyglucose–positronemission tomography (FDG-PET) and volumetric tumor assessments by CT/MRI.

#### 2.0 STUDY DESIGN

This phase 2, open-label, multicenter study will investigate the safety and efficacy of TAK-007 administered IV in adult patients with r/r B-cell NHL, including LBCL and iNHL, who have failed  $\geq 2$  prior systemic therapies. Eligible patients are required to have previously received an anti-CD20 monoclonal antibody (mAb) and chemotherapy regimen.

At the beginning of the study, the dose escalation phase will be conducted to assess the acute safety profile, CK, and pharmacodynamics of the TAK-007 cell product at 2 dose levels (200 × 106 [±30%] and 800 × 106 [±25%] CD19 CAR+ viable natural killer [NK] cells per patient). Previous clinical experience with CD19 CAR NK cells suggests that both proposed dose levels are likely to be clinically active [1]. A sequential dose escalation guided by Bayesian optimal interval (BOIN) design ([2], [3], [4]) will be used, followed by expansion cohorts to select the recommended phase 2 dose (RP2D).

#### 3.0 STATISTICAL HYPOTHESES AND DECISION RULES

### 3.1 Statistical Hypotheses

No longer applicable to the study as of Protocol Amendment 5.

#### 3.2 Multiplicity Adjustment

No longer applicable to the study as of Protocol Amendment 5.

### 4.0 SAMPLE-SIZE DETERMINATION

The primary analysis for the study does not involve any statistical inference. Consequently, the sample size was determined based on feasibility considerations instead of a formal statistical evaluation. Approximately 42 patients at dose levels of either  $200 \times 10^6$  (±30%) or  $800 \times 10^6$  (±25%) CD19-CAR+ viable NK cells per patient will be enrolled.

#### 5.0 ANALYSIS SETS

## 5.1 Intent-to-treat (ITT) Set

All enrolled patients in the TAK-007 study. This set will primarily be used for disposition.

# 5.2 Safety Analysis and Modified Intent-to-treat (mITT) Set

Patients who have received TAK-007 administration. This set will be used for safety analyses (safety set), and efficacy analysis to inform RP2D.

# 5.3 Response-Evaluable Analysis Set

Patients who have received TAK-007 administration, have had measurable disease at baseline, and at least 1 posttreatment radiologic assessment of disease response. This set will primarily be used for sensitivity analyses of efficacy endpoints, ORR and CR.

# 5.4 CK Analysis sets

CK Analysis Set (CKAS): All patients who have received TAK-007 administration and have at least 1 plasma sample obtained and analyzed.

CK Evaluable Population: All patients who have received TAK-007 administration and have a sufficient data to estimate 1 or more CK parameters.

Concertation analyses will be based on the CKAS.

#### 5.5 Pharmacodynamic Analysis Set

Patients from the safety analysis set who have a baseline and at least 1 postbaseline sample assessment, will be used for pharmacodynamics analyses.

## 5.6 Per-Protocol (PP) Set

The PP set will include all enrolled patients who do not have a major protocol violation. All decisions to exclude patients from the PP set will be made prior to the database lock.

#### 6.0 STATISTICAL ANALYSIS

#### **6.1** General Considerations

Baseline values are defined as the last observed value prior to the first dose of lymphodepleting chemotherapy unless specified otherwise.

All p-values reported will be 2-tailed (unless specified otherwise) and rounded to 3 decimal places prior to assessment of statistical significance.

Means and medians will be presented to 1 more decimal place than the recorded data. Standard deviations (SDs) will be presented to 2 more decimal places than the recorded data. Confidence intervals (CI)s intervals will be presented using the same number of decimal places as the parameter estimate.

Where applicable, variables will be summarized descriptively by study visit. For the categorical variables, the counts and proportions of each possible value will be tabulated by treatment group. The denominator for the proportion will be based on the number of subjects who provided non-missing responses to the categorical variable. For continuous variables, the number of subjects with non-missing values, mean, median, SD, minimum, and maximum values will be tabulated.

A windowing convention will be used to determine the analysis value for a given study visit for observed data analyses.

Screen failure subjects will be grouped and listed at the end.

The primary analysis will be conducted and documented in a clinical study report (CSR) after all dosed patients in the study have had the opportunity to be assessed for response and safety for at least 6 months after TAK-007 administration. Additional analyses may occur after the primary analyses have been completed. These additional analyses will be descriptive. The data cutoff for final analysis for the CSR addendum will be conducted after all dosed patients have had the opportunity to complete long-term follow-up or if the study has been terminated by the sponsor.

All the endpoints (by dose levels in dose escalation, and by disease cohorts and dose regimens in expansion cohorts) will be summarized separately, unless specified otherwise.

### **6.1.1** Definition of Study Visit Windows

All data will be categorized based on the scheduled visit at which they were collected unless otherwise specified. These visit designators are predefined values that appear as part of the visit tab in the electronic case report form (eCRF).

#### 6.1.2 Conventions for Missing/Partial Dates in Screening Visit

The following rules apply to dates recorded during the screening visits:

- If only the day-component is missing, the first day of the month will be used if the year and the month are the same as those for the first dose of lymphodepleting chemotherapy. Otherwise, the 15th of the month will be used.
- If only the year is present, and it is the same as the year of the first dose of lymphodepleting chemotherapy, the 15th of January will be used unless it is later than the first dose, in which case the date of the first of January will be used, unless other data indicate that the date is earlier.
- If only the year is present, and it is not the same as the year of the first dose of lymphodepleting chemotherapy, the 15th of June will be used, unless other data indicates that the date is earlier.

# 6.1.3 Conventions for Partial or Missing Adverse Event Dates

AEs with start dates that are completely or partially missing will be analyzed as follows:

- If month and year are known but day is missing:
  - If month and year are the same as month and year of TAK-007 infusion date, then impute to the TAK-007 infusion date.
  - If month and year are different than month and year of TAK-007 infusion date, then impute to first day of the month.
- If year is known but day and month are missing:
  - If year is same as year of TAK-007 infusion date, then TAK-007 infusion date will be used instead.
  - If year is different than year of TAK-007 infusion date, then 1<sup>st</sup> of January of the year will be imputed.
- If all are missing, then the start date is imputed with TAK-007 infusion date.

Imputing missing AE start date is mandatory. After the imputation, all imputed dates are checked against the stop dates to ensure the stop date does not occur before start date.

AEs with stop dates that are completely or partially missing will be analyzed as follows:

- If "ongoing" is checked, no imputation is necessary.
- If month and year are known but day is missing, the last day of the month will be imputed.
- If year is known, but day and month are missing:
  - If YYYY < year of TAK-007 infusion date, then 31st of December will be imputed.
  - If YYYY = year of TAK-007 infusion date, then 31st of December will be imputed.
  - If YYYY > year of TAK-007 infusion date, then 1st of January will be imputed.
- If all are missing, then impute date to 31st of December, in the year of TAK-007 infusion.

After the imputation, all imputed dates are checked against the start dates to ensure the stop date does not occur before start date. If the imputed stop date occurs prior to start date, then keep the imputed date the same as the start date. If subject dies, then use death date for AE stop date.

## 6.1.4 Conventions for Missing Concomitant Medication/Therapy Dates

Concomitant medications/therapies with start dates that are completely or partially missing will be analyzed as follows:

- If month and year are known, but day is missing, then impute day to first of the month.
- If year is known, but day and month are missing, then 1st of January of the year will be imputed.
- If all is missing, then impute date to date of birth (DOB).
- If DOB is not available but age is available, then estimate DOB by using screening date and age (age = screening date DOB).

Concomitant therapies with stop dates that are completely or partially missing will be analyzed as follows:

- If "ongoing" is checked, no imputation is necessary
- If month and year are known but day is missing, the last day of the month will be imputed.
- If year is known, but day and month are missing:
  - If YYYY < year of TAK-007 infusion date, then 31st of December will be imputed.
  - If YYYY = year of TAK-007 infusion date, then 31st of December will be imputed.
  - If YYYY > year of TAK-007 infusion date, then 1st of January will be imputed.
- If all is missing, then impute date to 31st of December in the year of TAK-007 infusion.

Imputing missing concomitant therapies is optional. However, if it is to be done, the rules are outlined above. If a subject dies, the death date will be used for the concomitant therapies stop date. After the imputation, all imputed dates will be checked against the start dates to ensure stop date did not occur before start date. If the imputed stop date occurs prior to start date, then the imputed date will be the same as the start date.

# 6.1.5 Conventions for Partial or Missing Subsequent Medication/Therapy Dates

Subsequent therapies with start dates that are completely or partially missing will be analyzed as follows:

- When month and year are present and the day of the month is missing:
  - If the onset month and year are the same as the month and year of TAK-007 infusion date, the day of TAK-007 infusion date + 1 will be imputed.
  - If the onset month and year are not the same as the month and year of TAK-007 infusion date, the first day of the month will be imputed.

- When only a year is present:
  - If the onset year is the same as the year of TAK-007 infusion date, the date of TAK-007 infusion date + 1 will be imputed.
  - If the onset year is not the same as the year of TAK-007 infusion date, the first day of the year is imputed.
- If no components of the onset date are present, the date of TAK-007 infusion date + 1 will be imputed.

#### 6.1.6 Conventions for Partial or Missing Death Dates

- If death year and month are available, but day is missing:
  - If the year and month for the last date known to be alive are the same as the year and month of death date, death date will be the day after the last date known to be alive.
  - If the year and month for the last date known to be alive is earlier than the death date, death date will be the first day of the death month.
- If both month and day are missing for death date or a death date is completely missing, do not impute, and censor the subject survival time at the last date known to be alive.

## 6.2 Disposition of Subjects

The number of subjects screened, enrolled, treated with lymphodepleting chemotherapy and treated with TAK-007 will be summarized. The number of subjects in each analysis set will be provided. The reasons for discontinuing treatment and discontinuing study will also be summarized.

The summary will be presented by dose levels, by disease cohorts, and overall for the study.

The percentages will be based on the number of patients in the ITT population, except for the number of subjects screened.

For the screening phase, the clinical eligibility criteria that were not met by patients will also be tabulated. The number of subjects enrolled by country and site will also be summarized.

# 6.3 Demographic and Other Baseline Characteristics

# 6.3.1 Demographics and Baseline Characteristics

Demographics will be summarized by dose levels, by disease cohorts, and overall for the study using the ITT and mITT populations. Baseline demographic data to be evaluated will include age, sex, race, ethnicity, height, weight, and other parameters, as appropriate. Age will be calculated from date of birth to date of informed consent.

Throughout this study, baseline assessments are defined as those performed at the closest time on or prior to the start of lymphodepleting chemotherapy, unless specified otherwise.

Disease characteristics will also be summarized in a similar fashion including disease diagnosis at initial diagnosis and study entry, follicular lymphoma international prognostic index (FLIPI) score (FL only) at study entry, international prognostic index for diffuse large B-cell lymphoma (IPI, LBCL only) at study entry, progression of disease within 24 months of starting induction chemoimmunotherapy (POD24) (iNHL only), molecular classification status (ABC or GCB) at study (LBCL only), bone marrow involvement at initial diagnosis and study entry, extranodal involvement at initial diagnosis and study entry, Ann Arbor stage at initial diagnosis and study entry, and baseline Eastern Cooperative Oncology Group (ECOG) status. Time since initial diagnosis will also be summarized.

Continuous variables will be summarized by means, medians, standard deviations, and ranges; categorical variables will be summarized by counts and percentages. Other variables may also be included in this analysis by categorizing the continuous variables or re-categorizing existing categorical variables.

# 6.4 Medical History and Concomitant Medications

Medical history and concomitant medications will be analyzed in the ITT analysis set. A general medical history will be listed for all patients, with medical history defined as any start date prior to informed consent.

Concomitant medications will be coded by generic term using the World Health Organization (WHO) Drug Dictionary. The number and percentage of patients taking concomitant medications from screening through the end of the on-study period will be tabulated by Anatomical Therapeutic Chemical (ATC) classification pharmacological subgroup and WHO generic drug term and sorted in decreasing frequency based on the number of reports. A patient who has been administered several medications with the same preferred medication name will be counted only once. The preferred medication name will be used.

#### 6.5 Any Prior Interventions

# 6.5.1 Prior Anti-cancer Therapy

Types of prior anticancer therapy will be summarized by dose levels, by disease cohorts and overall, along with number of lines, and best response to the most recent anticancer chemotherapy.

The status of refractory and relapsed as the response to last line of therapy, status of refractory and sensitive as the response to last line of chemotherapy, treatment history (primary refractory disease or never in CR) will also be summarized.

#### 6.5.2 Other Prior Interventions

A listing of prior surgery or procedure will be provided.

Types of prior radiotherapy and best response to the most recent prior radiotherapy will be summarized.

Types of prior stem cell transplant and source of stem cells will also be summarized.

#### 6.6 Efficacy Analysis

The mITT set will be used to inform the RP2D. The analyses of primary and secondary endpoints will be summarized by dose levels in the dose escalation cohorts, and by disease cohorts and dose regimens in expansion cohorts.

In the event a patient undergoes a stem cell transplantation (SCT) or any other anticancer therapy (excluding localized radiotherapy and surgery) while on study, the patient's best response will be derived only based on evaluation before SCT or initiation of a new therapy, whichever occurs earlier. All patients who do not meet the criteria for an objective response by the analysis cutoff date will be considered non-responders within the response-related analyses.

#### 6.6.1 Primary Endpoint Analysis

No longer applicable to the study as of Protocol Amendment 5.

# 6.6.2 Secondary Efficacy Endpoint(s) Analysis

#### 6.6.2.1 ORR by Investigator

ORR by investigator will be calculated by dose levels in the dose escalation cohorts, and by disease cohorts and dose regimens in expansion cohorts. 95% exact CI will be provided.

The subject incidence of best response (CR, partial response [PR], stable disease, progressive disease [PD]) by investigator will also be calculated, along with the 95% exact CI.

# 6.6.2.2 CR by Investigator

CR rate is defined as the incidence of CR as best response to treatment. CR by investigator will be presented along with the calculated 95% CI based on the binomial distribution.

# 6.6.2.3 DOR by Investigator

DOR is defined only for patients who experience objective response (CR or PR) and is the time from the date of first documented objective response to the date of first documented disease progression or death, whichever comes first. Patients not meeting the criteria for progression or death will be censored at the last disease assessment. Duration of response will be derived using disease assessments obtained on study prior to initiation of new anticancer therapy. Detailed handling rules for missing assessments and censoring for the analysis of DOR are presented in Table 1.

Table 1 Handling of Missing Assessments and Censoring for DOR Primary Analysis

| Situation | Date of progression or censoring | Outcome |
|---|---|---|
| PD documented at a scheduled visit or<br>between scheduled visits prior to<br>initiation of new anticancer therapy | Date of progression | Event |

| PD or death documented after at least | Date of last adequate assessment <sup>a</sup> | Censored |
|---|---|---|
| two missing tumor assessments | | |
| New anticancer therapy (excluding SCT | Date of last adequate assessment prior | Censored |
| and localized radiotherapy/surgery) started before documented progression or death | to initiation of anticancer therapy (excluding SCT and localized radiotherapy/surgery) | Lekins, |
| SCT started before documented progression or death | Date of SCT | Censored |
| No documented PD or death | Date of last adequate assessment | Censored |
| Lost to follow-up or withdrawal of consent | Date of last adequate assessment | Censored |

<sup>&</sup>lt;sup>a</sup> The date of the last assessment with response assessment as CR, PR or stable disease which was made before a censoring reason occurred.

Kaplan-Meier plots, estimates and median values (if estimable) along with their 2-sided 95% CIs, will be computed. Estimates of the proportion of event-free patients at 3-month intervals will be provided.

# 6.6.2.3.1 Sensitivity Analysis

Additional sensitivity analyses may also be performed based on the alternations of the handling of missing assessment and censoring in Table 2, on the basis of 1 alteration at a time, not on combined alterations unless otherwise specified. A sensitivity analysis combing the first 2 rows in Table 2 may also be conducted.

Table 2 Handling of Missing Assessments and Censoring for DOR Sensitivity Analysis

| Situation | Date of progression or censoring | Outcome |
|---|---|---|
| PD or death documented after at least two missing tumor assessments | Date of progression or death | Event |
| New anticancer therapy started before documented progression or death | Date of documented disease progression or death | Event |
| PD documented between scheduled visits prior to initiation of new anticancer therapy | Date of next scheduled assessment | Event |
| New anticancer therapy started before documented progression or death | Date of initiation of anticancer therapy | Censored |

## 6.6.2.4 PFS by Investigator

PFS in the mITT set is defined as the time from TAK-007 administration to the date of disease progression or death from any cause, whichever comes first. PFS in the ITT set is defined as the time from enrollment to the date of disease progression or death from any cause, whichever comes first. Patients who do not have disease progression or die will be censored at the last disease assessment. Patients who do not have postbaseline disease assessment prior to new anticancer therapy in the absence of death will be censored at the date of TAK-007 administration (mITT set) or enrollment (ITT set). Detailed handling rules for missing assessments and censoring will follow Table 1. Sensitivity analysis may be performed following censoring rules similarly as defined in Section 6.6.2.3.1.

Kaplan-Meier plots, estimates, and median values (if estimable) along with their 2-sided 95% CIs, will be computed. Estimates of the proportion of event-free patients at 3-month intervals will be provided.

#### 6.6.2.5 OS

OS in the mITT set is defined as the time from TAK-007 administration to the date of death. OS in the ITT set is defined as the time from enrollment to the date of death. Patients who do not die will be censored at the last contact date.

Kaplan-Meier plots, estimates and median values (if estimable) along with their 2-sided 95% CIs, will be computed. Estimates of the proportion of event-free patients at 3-month intervals will be provided.

# **6.6.3 Subgroup Analyses**

Subgroup analyses of the primary endpoint is no longer applicable with Protocol Amendment 5. Subgroup analyses may be performed for secondary endpoints CR, DOR, PFS and OS, if deemed appropriate.

The following baseline covariates may be used in the subgroup analyses. Subgroup analysis may also be performed in FL patients only.

- Gender: male, female
- Age at baseline:  $<65, \ge 65; <75, \ge 75 \text{ years}$
- Disease type in LBCL cohort: High grade B cell lymphoma, diffuse large B-cell lymphoma (DLBCL)-not otherwise specified (NOS), transformed DLBCL, primary mediastinal B cell lymphoma (PMBCL), others
- Disease type in iNHL cohort: FL, marginal zone lymphoma (MZL), subtypes of MZL (extranodal MZL, nodal MZL, splenic MZL)
- Response to last line of therapy: refractory, relapsed

- Refractory is defined as patients who experienced disease progression as best response
  to last line of therapy or had stable disease after last line of therapy with duration of
  stable disease no longer than 6 months.
- Relapsed is defined as patients who had a CR or PR from last line of prior therapy and relapsed prior to the study.
- Response to last line of chemotherapy: refractory, sensitive
  - Refractory is defined as patients who never achieved CR or PR after the last line of chemotherapy.
  - Sensitive is defined as patients who achieved CR or PR after the last line of chemotherapy.
- Treatment history: primary refractory disease, never in CR
  - o Primary refractory is defined as patients who experienced disease progression as best response to first line therapy or had stable disease after the first line therapy with duration of stable disease no longer than 6 months from the last dose of therapy.
  - o Never in CR is defined as patients who never achieved CR to any line of prior therapy.
- Prior autologous stem cell transplantation: Yes, No
- Prior allogeneic stem cell transplantation: Yes, No
- Type of Prior CD19 therapy: CD19 Targeted Therapy, CD19 CAR-T, CD19 T-Cell Engager
- Number of prior lines of systemic treatment:  $2, \ge 3$
- Disease stage at study entry: 1 or II, III or IV
- Disease stage at initial diagnosis: I or II, III or IV
- LBCL cohort:
  - o IPI risk category at study entry: 0-2, 3-5
  - IPI risk category at initial diagnosis: 0-2, 3-5
- FL cohort
  - FLIPI score at study entry: 0-2, 3-5
  - FLIPI score at initial diagnosis: 0-2, 3-5
- History of bone marrow involvement: Yes, No
- Tumor burden by metabolic tumor volume at baseline: ≤median, >median
- Lactate dehydrogenase (LDH) at baseline: <500 U/L, ≥500 U/L
- Extranodal disease at baseline: Yes, No
- Beta-2 microglobulin: ≤3 mg/L, >3 mg/L

- Cell of origin in LBCL cohort: germinal center B-cell-like subtype, activated B-cell-like subtype
- Rearranged MYC plus BCL2, BCL6 or both in LBCL cohort: double or triple hit, not double
  or triple hit
- POD24 in iNHL cohort: Yes, No
  - o POD24 is defined as disease progression within 24 months from the start of systemic chemo-immunotherapy or during CD20 mAb maintenance.
- Time to progression in LBCL cohort: <12 month, <24 month and ≥12 month, ≥24 month
  - Time to progression is defined as time between start of first-line chemo-immunotherapy treatment until first disease progression.
- PRIMA-PI score for FL at study entry: high-risk, intermediate-risk, low-risk
  - O High-risk is defined as Beta-2 microglobulin > 3 mg/L
  - o Intermediate-risk is defined as Beta-2 microglobulin ≤ 3mg/L with bone marrow involvement at baseline
  - Low-risk is defined as Beta-2 microglobulin ≤ 3mg/L without bone marrow involvement at baseline

#### 6.7 Safety Analysis

#### **6.7.1** Adverse Events

The safety set will be used for all safety analyses.

Treatment-emergent adverse events (TEAE) are defined as any AE that begins on or after the start date of lymphodepleting chemotherapy.

The incidence and percentages of TEAEs will be summarized by System Organ Class (SOC) and Preferred Term (PT) of the International Council for Harmonisation Medical Dictionary for Regulatory Activities (MedDRA) and by grade according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 [5]. In addition, grading of cytokine release syndrome (CRS) and immune effector cell-associated neurotoxicity syndrome (ICANS) will follow the American Society for Transplantation and Cellular Therapy (ASTCT) guidelines [6], grading of acute graft-versus-host disease (GvHD) will follow the recommendations by the Mount Sinai Acute GvHD International Consortium [7], and grading of chronic GvHD will follow the 2014 National Institutes of Health (NIH) Consensus [8]. For each set of grading criteria, a later version of the criteria may be applied.

Tabulated AEs will include the following categories:

- TEAEs.
- Grade >3 TEAEs.
- Grade  $\geq 3$  drug-related TEAEs.
- The most commonly reported TEAEs (ie, those events reported by ≥10% of patients).

  Serious adverse events (SAEs).

  Drug-related SAEs.

  Deaths.

- Drug-related deaths.
- Adverse events of clinical interest (AECIs) as defined in Section 6.7.2.

Additionally, any TEAE leading to treatment discontinuation (lymphodepleting chemotherapy or TAK-007) will be summarized. A listing will be provided.

AEs that begin on or after the date of signed informed consent but before the start date of lymphodepleting chemotherapy will be provided in a listing.

#### **Adverse Events of Clinical Interest** 6.7.2

The sponsor has designated some AEs as being of clinical interest. Since there are no commercially available CAR-NK therapies, TEAEs of clinical interest are based on adverse reactions reported with commercially available CAR-T therapies and common adverse reactions related to lymphodepleting chemotherapy. Rates of all AECIs are expected to be lower in patients treated with TAK-007 compared to rates in patients treated with CAR-T therapies. AECIs related to lymphodepleting chemotherapy are expected to have comparable rates to those described in the cyclophosphamide and fludarabine product labeling.

The list of AECIs includes:

- CRS:
  - Hemophagocytic lymphohistiocytosis (HLH)
  - Macrophage activation syndrome (MAS)
- ICANS (including encephalopathy, seizures, confusion, somnolence, aphasia, and cerebral edema)
- Tumor lysis syndrome (TLS)
- Hypersensitivity reactions/Infusions reactions
- Myelosuppression (including neutropenia, opportunistic infections, thrombocytopenia, bleeding, and anemia)
- Second primary malignancies

These TEAEs of clinical interest are defined using Standardised MedDRA Queries (SMQs),

The analyses of TEAEs of clinical interest will be conducted using the safety analysis set, as similar fashion described in Section 6.7.1.

#### 6.7.3 **Other Safety Analysis**

Descriptive statistics for the actual values of clinical laboratory parameters will be presented for all scheduled measurements over time. Mean laboratory values over time will be plotted for key laboratory parameters. Shift tables for laboratory parameters will be generated for changes in NCI CTCAE grade from baseline to worst postbaseline value.

Descriptive statistics for the actual values (and/or the changes from baseline) of vital signs and electrocardiograms (ECGs) will be tabulated by scheduled time point. ECOG performance scores will also be summarized using shift tables.

#### 6.7.4 **Extent of Exposure and Compliance**

The exposure to fludarabine and cyclophosphamide will be characterized by total amount of dose received (mg), total number of doses received, and relative dose intensity using safety set. The number and percentage of patients whose dose was modified or discontinued will be summarized.

The relative dose intensity (%) is defined as:  $100 \times (\text{total dose received})/(\text{total dose intended})$ . Total dose intended is the summation of the intended doses on Days -5, -4 and -3.

The exposure to TAK-007 will be characterized by total number of NK cells in prepared product, total number and percentage of transduced CAR+ cells in prepared product, total number of NK cells infused to patients, total number and percentage of transduced CAR+ cells infused to patients, and viability in the prepared product using safety set.

The exposure will be summarized separately by dose levels and disease indications.

#### 6.8 CK, Pharmacodynamic, and Other Analyses

#### 6.8.1 **CK Analyses**

#### CK Sample Collection and Analysis:

Blood samples will be collected at pre-dose and 1 hour (±15 minutes) after TAK-007 administration on Day 0, Day 1, Day 3, Day 5, Day 7, Day 10, Day 14, Day 21, Day 28/Month 1, Month 2, Month 3, Month 4 and Month 6 for primary analysis and analyzed for TAK-007 transgene copies per genomic DNA by Droplet Digital Polymerase Chain Reaction (ddPCR) and TAK-007 CAR+ NK cell number by flow cytometry.

#### **Summary Statistics:**

Individual blood level of TAK-007 (as transgene copies per genomic DNA) and TAK-007 cell number (as CAR+ NK cells/µL) versus time data will be listed by dose level or indication. Individual blood level of TAK-007 and TAK-007 cell number versus actual time profiles will be plotted on both linear and semi logarithmic scales for each subject. Blood levels of TAK-007 and TAK-007 cell number will be summarized by nominal time point for each dose level and indication using the following descriptive statistics includes n, arithmetic mean, SD, percent coefficient of variation (CV%), median, minimum and maximum. Blood level of TAK-007 and TAK-007 cell numbers will be reported to 3 significant figures in summary statistics except for CV% which will be reported to 1 decimal place. Sample side (N) will be presented as an integer.

Blood level of TAK-007 and TAK-007 cell number concentrations that are below the limit of quantification (BLQ) will be set to zero for calculation of summary statistics.

# Noncompartmental Analysis:

CK parameters will be estimated using noncompartmental methods by Phoenix® WinNonlin® (Certara L.P., Princeton, NJ) Version 8.0 or higher. In addition, separate population-based CK analysis may be performed using NONMEM 7 (ICON plc, Dublin, Ireland). The actual sampling and dose duration times will be used for the calculation of CK parameters.

As permitted by data, CK parameters will be estimated from the blood level of TAK-007 and TAK-007 cell number versus time profiles using the CK analysis set as the following.

| CK Parameter | Definition |
|---|---|
| $C_{max}$ | Maximum observed concentration |
| $T_{\text{max}}$ | Time to maximum observed concentration |
| AUC <sub>last</sub> | Area under the concentration versus time curve (AUC) from time 0 to the last |
| | quantifiable measurement, calculated using the linear trapezoidal rule |
| $AUC_{(0-28)}$ | AUC from time 0 to Day 28 post dose |
| AUC <sub>(0-90)</sub> | AUC from time 0 to Month 3 post dose |
| $C_{28}$ | Concentration at Day 28 |
| C <sub>last</sub> | The last quantifiable measurement |
| T <sub>last</sub> | The last quantifiable time point |

Table 3 Cellular Kinetic Parameters Estimated Using Noncompartmental Analysis

For the calculation of CK parameters, all BLQ will set to missing except that prior to the first measurable value will be set to zero. The BLQ values that are between measurable values will be set to missing

If a patient deviated substantially from the protocol-defined study procedures, including but not limited to dosing, dose timing, sample collection, and concomitant medications, CK parameters will be included in the listings but excluded from the descriptive statistics and statistical evaluations, with appropriate footnotes.

Individual CK parameters will be listed and also summarized as permitted by data by part, cohort and indication using descriptive statistics: the n, arithmetic mean, SD, CV%, minimum, median, maximum, and geometric mean and geometric CV%. T<sub>max</sub> will be summarized by n, minimum, median, and maximum only.

CK parameters will be reported to 3 significant figures in summary statistics except for CV% and geometric CV%, which will be reported to 1 decimal place.

Descriptions of population CK modeling methods and data analysis will be documented and reported in a separate brief report.

# 6.8.2 Pharmacodynamic Analyses

Changes in average B cell counts from baseline will be summarized. The frequency and percentage of patients with B cell aplasia will be summarized before and after TAK-007 administration by scheduled time point using the pharmacodynamic analysis set. B cell aplasia is defined as <50 B cell/ul of blood

Concentration data of interleukin (IL)-15 and soluble immune factors in circulation (eg, interferon gamma, IL-1 $\beta$ , IL-2, IL-4, IL-6, IL-10, IL-12p70, IL-13, tumor necrosis factor alpha, granulocyte-macrophage colony-stimulating factor) in plasma will be tabulated using summary statistics over scheduled time point. Individual and mean concentration-time profiles may also be plotted.

Additional analysis may be performed as appropriate and will be reported outside the CSR.

#### 6.9 Immunogenicity Analyses

Frequency and percentage of patients with detectable anti-HLA (including donor specific anti-HLA antibodies) and anti-CAR antibodies will be summarized by scheduled time point using the safety analysis set. Impact of anti-HLA and anti-CAR immunogenicity on CK parameters, safety and efficacy may be assessed, as appropriate based on the available data.

#### 6.10 RCR Analyses

Frequency and percentage of patients with positive RCR test results will be summarized by scheduled time point before and after TAK-007 administration using safety analysis set.

# 6.11 Exploratory Analyses

#### 6.11.1 Population CK-Pharmacodynamic Analysis

The relationship between TAK-007 systemic exposure and safety, efficacy, and pharmacodynamic response (eg, B cell aplasia, time to B cell recovery, changes in cytokines/chemokines) will be evaluated to understand the CK-pharmacodynamic relationship of TAK-007. These data will be reported outside the CSR.

#### **6.11.2** Biomarker Analyses

Exploratory biomarker analyses will be separately defined in biomarker analysis plan and the results of these analyses may be reported separately from the CSR.

#### 6.11.3 **Imaging Analyses**

As data permit, the metabolic tumor volume measures including standard uptake value, lesion Analyses to understand the relationship between metabolic tumor volume and patients response may be evaluated. volumes and total lesion glycolysis as assessed by FDG-PET will be summarized at baseline. 

#### 6.11.4 **Patient-Reported Outcome Analyses**

No longer applicable to the study as of Protocol Amendment 5.

#### 6.11.5 **Healthcare Resource Utilization Analyses**

No longer applicable to the study as of Protocol Amendment 5.

#### 6.12 **Statistical Considerations for Dose Escalation**

A sequential dose escalation guided by BOIN design ([2], [3], [4]) will be used followed by expansion cohorts to select the RP2D.

During the dose escalation, only patients who received TAK-007 will be considered as doselimiting toxicity (DLT)-evaluable. Each dose level will enroll at least 3 patients. The target toxicity rate for the maximum tolerated dose (MTD) is  $\phi = 0.25$ , and the maximum sample size is 12 total patients for dose escalation. As shown in Table 4, the BOIN design uses the following rule to guide dose escalation/ de-escalation:

- If the observed DLT rate at the current dose is  $\leq 0.197$ , escalate the dose to the next higher dose level; if the current dose is the highest dose, treat the new patients at the highest dose.
- If the observed DLT rate at the current dose is > 0.298, de-escalate the dose to the next lower dose level; if the current dose is the lowest dose and the rule indicates dose deescalation, treat the new patients at the lowest dose unless the number of DLTs reaches the elimination boundary (as shown in Table 4), at which point the dose escalation will be terminated for safety.
- Otherwise, stay at the current dose.
- Repeat above until the maximum sample size of 12 is reached, or until the number of evaluable patients treated at the current dose reaches 6 and the decision according to above is to stay at the current dose.

For the purpose of overdose control, doses i and higher levels will be eliminated from further examination if  $Pr(p \neq 0.25 \mid data) > 0.95$  and at least 3 evaluable patients have been treated at dose level j, where p j is the true DLT rate of dose level j, j=1, 2.

Table 4 Dose Escalation/De-escalation Rule for the BOIN Design

| Number of Evaluable Patients<br>Treated at Current Dose | 1 | 2 | 3 | 4 | 5 | 6 |
|---|---|---|---|---|---|---|
| Escalate if # of DLT ≤ | 0 | 0 | 0 | 0 | 0 | 1 |
| De-escalate if # of DLT ≥ | 1 | 1 | 1 | 2 | 2 | 2 |
| Eliminate if # of DLT $\geq$ | NA | NA | 3 | 3 | 3 | 4 / 2 |

DLT: dose-limiting toxicity

"# of DLT" is the number of patients with at least 1 DLT. When none of the actions (i.e., escalate, de-escalate or eliminate) is triggered, stay at the current dose for treating the next cohort of patients. "NA" means that a dose cannot be eliminated before treating 3 evaluable patients.

Enrollment into the lower dose level may be continued during exploration of the higher dose level in the dose escalation phase, if deemed appropriate by the sponsor and the investigators. In this case, if additional DLT are identified during additional patients enrolled, the dose escalation decision will be re-examined using the cumulative DLT rate at this dose level.

Separate expansion cohorts for LBCL and iNHL with approximately 15 patients each may be initiated for dose level(s) selected based on the dose escalation part, to further evaluate the safety, tolerability, efficacy and cellular kinetics and allow the selection of the RP2D to be used in the rest of the study.

# 6.13 Interim Analysis and Criteria for Early Termination

No longer applicable to the study as of Protocol Amendment 5.

#### 6.14 Data Monitoring Committee

No longer applicable to the study as of Protocol Amendment 5.

# 7.0 REFERENCES

- Liu, E., Marin, D., Banerjee, P., Macapinlac, H. A., Thompson, P., Basar, R., et al. 2020. Use of CAR-Transduced Natural Killer Cells in CD19-Positive Lymphoid Tumors. N Engl J Med, 382(6), 545-53.
- 2. Liu S, Yuan Y. Bayesian Optimal Interval Designs for Phase I Clinical Trials. J R Stat Soc Ser C Appl Stat 2015;64(3):507-23.
- 3. Yuan Y, Hess KR, Hilsenbeck SG, Gilbert MR. Bayesian optimal interval design: A simple and well-performing design for phase i oncology trials. Clin Cancer Res 2016;22(17):4291-301.
- 4. Zhou, H., Yuan, Y., & Nie, L. (2018). Accuracy, safety, and reliability of novel phase I trial designs. Clinical Cancer Research, 24(18), 4357-4364.

- 5. Common Terminology Criteria for Adverse Events (CTCAE). National Cancer Institute, National Institutes of Health, U.S. Department of Health and Human Services Series v 5.0. 27 November 2017.
- 6. Lee, D. W., Santomasso, B. D., Locke, F. L., Ghobadi, A., Turtle, C. J., Brudno, J. N., et al. 2019. ASTCT consensus grading for cytokine release syndrome and neurologic toxicity associated with immune effector cells. *Biol Blood Marrow Transplant*, 25(4), 625-38.
- 7. Harris AC, Young R, Devine S, Hogan WJ, Ayuk F, Bunworasate U, et al. International, multicenter standardization of acute graft-versus-host disease clinical data collection: a report from the Mount Sinai GVHD international Consortium. Biol Blood Marrow Transplant. 2016; 22(1):4-10.
- 8. Jagasia MH, Greinix HT, Arora M, Williams KM, Wolff D, Cowen EW, et al. National Institutes of Health consensus development project on criteria for clinical trials in chronic graft-versus-host disease: I. The 2014 diagnosis and staging working group report. Biol Blood Marrow Transplant. 2015; 21(3): 389-401.

# 8.0 CHANGES TO PROTOCOL PLANNED ANALYSES

NA

#### 9.0 APPENDIX

SAS version 9.4 or higher will be used for the analysis.

# 10.0 CHANGES FROM THE PREVIOUS VERSION OF THE SAP

| SAP Section | Impacted Text (shown in bold) | Change | Rationale for Change |
|---|---|---|---|
| 1.0 OBJECTIVES AND ENDPOINTS | or, | Removed all objectives and endpoints associated with Part 2 of the study. | Part 2 of the study was removed with protocol amendment 5. |
| 2.0 STUDY DESIGN | | Removed portion which summarized design for Part 2. | Part 2 of the study was removed with protocol amendment 5. |
| 3.0 STATISTICAL<br>HYPOTHESIS AND<br>DECISION RULES | | Removed this section as<br>the study no longer has a<br>formal hypothesis with<br>the removal of Part 2. | Part 2 of the study was removed with protocol amendment 5. |
| 4.0 SAMPLE-SIZE<br>DETERMINATION | The primary analysis for the study does not involve any statistical inference. Consequently, the sample size was determined based on feasibility considerations instead of a formal | Removed the calculation<br>for Part 2 and included<br>additional details around<br>the primary analysis. | Part 2 of the study was removed with protocol amendment 5. |

| | statistical evaluation. Approximately 42 patients at dose levels of either 200 × 10 <sup>6</sup> (±30%) or 800 × 10 <sup>6</sup> (±25%) CD19-CAR+ viable NK cells per patient will be enrolled. | | ide Terms of |
|---|---|---|---|
| 5.4 CK ANALYSIS SET | CK Analysis Set (CKAS): All patients who have received TAK- 007 administration and have at least 1 plasma sample obtained and analyzed. CK Evaluable Population: All patients who have received TAK- 007 administration and have a sufficient data to estimate 1 or more CK parameters. | Provided additional details about the CK analysis sets | More clearly define the CK populations |
| 6.1 General<br>Considerations | The primary analysis will be conducted and documented in a clinical study report (CSR) after all dosed patients in the study have had the opportunity to be assessed for response and safety for at least 6 months after TAK-007 administration. AEs with start dates that are completely or partially missing will be analyzed as follows: | Updated language to correct use of acronyms | Align this section with the rest of the document |
| 6.2 Disposition of<br>Subjects | | Removed mention of Part 2. | Part 2 of the study was removed with protocol amendment 5. |
| 6.3 Demographics and<br>Other Baseline<br>Characteristics | | Removed mention of Part 2. | Part 2 of the study was removed with protocol amendment 5. |
| 6.6 Efficacy Analysis | | Removed analyses associated with Part 2. | Part 2 of the study was removed with protocol amendment 5. |
| 6.6 Efficacy Analysis | In the event a patient<br>undergoes a stem cell<br>transplantation (SCT) or | Included additional details that subjects will not be censored at localized | Patients will not be<br>censored if they received<br>anticancer therapy which |

| | any other anticancer<br>therapy (excluding<br>localized radiotherapy<br>and surgery) while on<br>study | radiotherapy or surgery. | is deemed to not affect the disease of interest. |
|---|---|---|---|
| 6.6.3 Subgroup Analyses | • Type of Prior CD19<br>therapy: CD19 Targeted<br>Therapy, CD19 CAR-T,<br>CD19 T-Cell Engager | Included additional<br>subgroup around type of<br>Prior CD19 therapy | Me Lekins |
| 6.7 Safety Analysis | | Removed mention of Part 2. | Part 2 of the study was removed with protocol amendment 5. |
| 6.7.1 Adverse Events | | Removed summaries<br>specific to the time<br>between lymphodepleting<br>chemotherapy and TAK-<br>007 Administration, and<br>solely after TAK-007<br>administration | 2 |
| 6.8.1 CK Analyses | If a patient deviated substantially from the protocol-defined study procedures, including but not limited to dosing, dose timing, sample collection, and concomitant medications, CK parameters will be included in the listings but excluded from the descriptive statistics and statistical evaluations, with appropriate footnotes. | Updated analyses to align with protocol amendment 5 | |
| 6.11 Exploratory Analysis | | Removed analysis of<br>Time to Next Therapy | Align with protocol amendment 5 |
| 6.11.4 Patient-Reported<br>Outcome Analyses | | Removed all PRO<br>Analyses as these were<br>specific to Part 2. | Part 2 of the study was removed with protocol amendment 5. |
| 6.11.5 Healthcare<br>Resource Utilization<br>Analyses | | Removed all healthcare resource utilization analyses as these were specific to Part 2. | Part 2 of the study was removed with protocol amendment 5. |
| 6.13 Interim Analysis and<br>Criteria For Early<br>Termination | | Removed as the interim analysis was specific to Part 2. | Part 2 of the study was removed with protocol amendment 5. |
| 6.14 Data Monitoring<br>Committee | | Removed as the DMC was specific to Part 2. | Part 2 was removed with protocol amendment 5. |

Protety of Takeda. For noncommercial use only and subject to the applicable Terms of use

# Signature Page for 16-1-9-1 Statistical Analysis Plan 2024-08-30 Title: TAK-007-2001 Statistical Analysis Plan 2024-08-30

| Title: TAK-007-2001 Statistical Analysis Plan 2024-08-30 | | , Jse |
|---|---|---|
| Approval | Statistics<br>04-Sep-2024 16:13:08 GMT+0000 | Letines of |

Property of Takeda: For non-commercial use only and subject to the admicable